CLINICAL TRIAL: NCT00035009
Title: A Double-Blind, Multicenter, Placebo- and Active-Controlled Acute and Extension Study of MK0869 in the Treatment of Patients With Major Depressive Disorder With Melancholic Features
Brief Title: Treatment of Patients With Major Depressive Disorder With MK0869 (0869-059)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0869-059; Formally-1A407; MK0869-059; 2006_402
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0869, aprepitant
Drug: Comparator: paroxetine HCL

SUMMARY:
A clinical study to determine the efficacy and safety of MK0869 in the treatment of depression

DETAILED DESCRIPTION:
The duration of treatment is 8 weeks.

ELIGIBILITY:
Major Depressive Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2001-09-20 (Actual); Primary Completion 2003-12-22 (Actual); Study Completion 2004-03-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HAMD-17 total score at week 8. Mk-0869 will be generally well tolerated

SECONDARY OUTCOMES:
Actual CGI-I score at week 8, improving social disability by change from baseline in Sheehan Disability Score at Week 8, change from baseline in the HAMA score at week 8, change from baseline in depressed mood of the HAMD-17 at week 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Liu KS, Snavely DB, Ball WA, Lines CR, Reines SA, Potter WZ. Is bigger better for depression trials? J Psychiatr Res. 2008 Jul;42(8):622-30. doi: 10.1016/j.jpsychires.2007.07.003. Epub 2007 Sep 7. PMID 17825841
- [Result] Keller M, Montgomery S, Ball W, Morrison M, Snavely D, Liu G, Hargreaves R, Hietala J, Lines C, Beebe K, Reines S. Lack of efficacy of the substance p (neurokinin1 receptor) antagonist aprepitant in the treatment of major depressive disorder. Biol Psychiatry. 2006 Feb 1;59(3):216-23. doi: 10.1016/j.biopsych.2005.07.013. Epub 2005 Oct 24. PMID 16248986
- Available data/document: CSR Synopsis Links — http://www.merck.com/clinical-trials/policies-perspectives.html